CLINICAL TRIAL: NCT00054730
Title: Effects of Ampakine CX516 (Ampalex®) on Functioning in Fragile X Syndrome and Autism
Brief Title: Effects of CX516 on Functioning in Fragile X Syndrome and Autism
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: RespireRx (Industry)
Collaborators: FRAXA Research Foundation (Other)
Organization: Cortex (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CORX-CX516-013
Record Dates: First submitted 2003-02-07; First posted 2003-02-11 (Estimated); Last update posted 2005-06-24 (Estimated); Status verified 2005-02

CONDITIONS: Fragile X Syndrome; Autism
Keywords: Fragile X Syndrome; Autism
MeSH Terms: conditions — Fragile X Syndrome; Autistic Disorder | interventions — 1-(quinoxalin-6-ylcarbonyl)piperidine

INTERVENTIONS:
Drug: CX516 (Ampalex®)

SUMMARY:
This study will investigate whether CX516 can improve attention, memory, language, or behavior in adults with Fragile X Syndrome and/or Autism.

CX516 is an AMPAKINE® compound. AMPAKINE compounds enhance synaptic strength. There is evidence to suggest that the synapses in the brain of an individual with fragile X syndrome are immature and abnormal. It is possible CX516 may partially correct this synaptic transmission defect and lead to improvement in cognitive and behavioral functioning.

There is also reason to believe that these changes caused by CX516 could be helpful in managing cognitive and behavioral symptoms in patients with autistic disorder.

Involvement for each participant will last 28 days. Participants will be given study medication, a physical exam, and a variety of cognitive assessment tests to study potential drug effectiveness at improving disease symptoms.

ELIGIBILITY:
Inclusion criteria:

Fragile X group

* DNA-based diagnosis of Fragile X syndrome

Autism group

* Documented diagnosis with ADOS; ADI-R; CARS and GARS

Both groups

* 18-50 years
* Measured IQ below 85
* Measured IQ >20
* Mental age >30 months
* Stable medication regimen for past 8 weeks
* Normal hearing
* Vision corrected to at least 20/50
* All females of childbearing age must have a negative pregnancy test at enrollment

Exclusion criteria:

* Recent history of seizure, epilepsy, or blackouts
* Unresolved medical issue impacting performance
* Behavioral dysfunction to the point that subject cannot cooperate for testing
* History of drug-induced neutropenia
* Uncontrolled hypertension

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Dates: Start 2002-06

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - UC Davis-MIND Institute, Sacramento, California
  - RUSH-Presbyterian-St. Luke's Medical Center, Chicago, Illinois

REFERENCES:
- See also: Fraxa is a research foundation whose mission is to support research aimed at treatment for Fragile X syndrome. — http://www.fraxa.org